CLINICAL TRIAL: NCT02769000
Title: Phase IIa Trial of Low Dose Radiation THerapy to Reduce Cerebral Amyloidosis in Early Alzheimer's Dementia
Brief Title: Low Dose RT to Reduce Cerebral Amyloidosis in Early Alzheimer's
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was suspended in March of 2020 due to COVID. Rather than reopen the study, the decision was made to terminate it in July of 2021.
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20004955
Record Dates: First submitted 2016-04-05; First posted 2016-05-11 (Estimated); Results first posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-11

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects 1-30 (Experimental): 15 subjects in each RT dose schedule 10 GY in 5 daily fractions 20 GY in 10 daily fractions
  Interventions: Radiation: 10 GY in 5 daily fractions; Radiation: 20 GY in 10 daily fractions

INTERVENTIONS:
Radiation: 10 GY in 5 daily fractions — Subjects 1-15 10 GY in 5 daily fractions
Radiation: 20 GY in 10 daily fractions — Subjects 16-30 20 GY in 10 daily fractions

SUMMARY:
Evaluate safety and toxicity/adverse events associated with delivery of low dose whole brain irradiation in patients with early Alzheimer's dementia according to the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria.. As a secondary goal it will establish whether or not the intervention with low dose whole brain irradiation stabilizes or decreases cerebral amyloid deposits and whether these correlate with the recognized progression of Alzheimer's dementia. The investigators will also collect information from the FDG and Amyvid® PET Scans to determine if there is any correlation between neurocognitive/quality of life scores and changes in amyloid plaque size, number and location.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is currently the 7th leading cause of death in the United States with approximately 5.9 million Americans living with the progressive and debilitating condition. AD predominantly affects older individuals as 86% of AD cases are in individuals 65 years of age and older. Further, approximately $172 billion of health care spending annually can be attributed to costs associated with AD care on top of the 11 million caregivers that provide care in unpaid capacities, such as family members, friends, etc.

In 1975, a cohort of nearly 2,800 people who were 65 years of age and free of dementia provided a basis for an incident study of dementia, as well as for Alzheimer's disease. This cohort was followed for almost 29 years and its sentinel findings included a significantly higher lifetime risk for both Alzheimer's and dementia in women compared to men. The estimated lifetime risk was nearly one in five for women compared to one in ten for men. In addition to the higher lifetime risk in women, expectancy of longer life and the aging of the "baby boomers" combined with improved healthcare is expected to increase the number of Americans who will reach 85 years of age or more. It is very clear that as the age increases, so does the incidence of Alzheimer's and other forms of dementia.

Between 2010 and 2050, it is expected that there will be a 30% increase in the number of individuals greater that 85 years of age. Although the absolute number may not appear to be significant, this increase of approximately 17 million people will challenge the healthcare system because of the cost associated with dealing various acute and chronic medical conditions including AD.

While other major causes of death continue to experience decline, those from AD continues to rise. In 1991, only approximately 14,000 death certificates recorded Alzheimer's disease as an underlying cause. In 2006, it was noted that there was an increase of approximately 46% in which Alzheimer's disease was listed as the direct cause of death. This is significant when compared to the present leading cause of death, heart disease, which decreased by 11% in the same time.

From a neurophysiological standpoint, what is known about Alzheimer's disease is that there appears to be a progressive process that is associated with the deposition of β Amyloid. This appears to have a triggering mechanism, which causes the phosphorylation of a TAU protein, which then leads to development neurofibrillary tangles (NFT), which are believed to be responsible for memory loss, especially short-term and other associated problems with Alzheimer's related dementia. It also appears that there may be a selective deposition of the β Amyloid in the hippocampus and the prefrontal regions, which are the major short-term memory regions of the brain.

Extensive research has been ongoing to try to find various ways in which the excess deposition of β Amyloid, the removal of excess β Amyloid, the initiation sequence that it is involved in with phosphorylated TAU and other selective processes can be altered in an effort to mitigate the devastating end term results. To date, there have been several trials, including a vaccine trial performed in Europe and in the United States, which seem to show that clearance of the β Amyloid is possible. However, there was not significant improvement in neurocognitive function (NCF), which led to the discontinuation of these trials.

This lack of improvement in NCF was believed to be secondary to the fact that the β Amyloid had already resulted in the phosphorylation of the TAU protein and development of NFT. Thus removal of the initiator was accomplished, but only after the end damage had developed. Then why consider irradiation?

The use of radiation in the treatment of non-oncologic human populations has enjoyed a long history and a more recent renaissance. It is now commonly used to prevent heterotopic bone formation and re-development of keloids or heterotrophic scars post-operatively. It has been shown in a randomized trial to effectively treat planter fasciitis and has been used in post-operative treatment of resected pterygium. It has been used in the treatment of Hidradenitis suppurativa, Duputryen's disease and Ledderhose's disease. These sites routinely are treated with low dose fractionated external beam irradiation, commonly in doses that ranging from 7 to 24 Gy.

The use of external irradiation has also been reported in the treatment of symptomatic systemic amyloidosis. In published peer reviewed articles treatment sites have include trachea-pulmonary, ocular, laryngeal and for use as a conditioning agent for autologous BMT in patients with systemic amyloidosis. These reports used external beam irradiation that ranged from 5.5 - 45 Gy and detail durable local control with these doses.

Because of this effect, a series of basic science experiments were initiated with genetically altered mice: the B6; Cg - Tg 85 Dbo/J over express amyloid and the B6; 129-Psen1tm1MpmTg over express both amyloid and TAU, making them prone to early Alzheimer's disease development.

Both single and fractionated CNS irradiation in a genetically altered mouse model were tested, and have shown similar results with reduction in amyloid plaque number, size and volume. Moreover, the fractionated studies the investigators have demonstrated statistically significant improvement in the treated mice using the Morris Water Maze Test when compared to control non-treated animals, an effect which held up whether the animals were adolescent, mature or aged (up to 18 months old).

The exact mechanism by which radiation therapy confers benefit in the Alzheimer's disease mouse model will be difficult to elucidate as the exact pathobiology of Alzheimer's disease is not known. Possible mechanisms include the following: reduction of β amyloid by reducing production or increasing clearance; reduction in Tau; induction of beneficial inflammatory mechanisms; induction or inhibition of heat shock proteins; altering cerebral microvasculature; and/or reversal of maladaptive neuroplasticity in the hippocampus. Investigations of these possible mechanisms are currently underway.

One of the complications related to studying Alzheimer's disease is the actual diagnosis. Unlike malignancies where a biopsy can be obtained, Alzheimer's disease is a diagnosis of exclusion or made at autopsy. While the Europeans have recently identified and agreed on CSF biomarkers for diagnosis of Alzheimer's disease, the investigators have not accepted that premise in the United States. At the present time, PET imaging which utilizes various compounds has been utilized to identify depositions of amyloid in the CNS. More recently, there is some suggestive evidence that a specific type of cataract may be seen in a high percentage of patients with Alzheimer's disease related to possible β Amyloid deposition in the lens region (29-30). Many rely on the NINCDS-ADRDA criteria for clinical diagnosis of Alzheimer's disease.

While it is a diagnosis of exclusion, there are well-accepted neurocognitive tests (NCT) used to monitor Alzheimer's disease progression. The Mini Mental exam is one of the general NCT used to help establish the diagnosis of Alzheimer's dementia. There are other more sensitive neurocognitive tests available to track progression of Alzheimer's dementia, which the investigators will use in this study. Note estimation of premorbid IQ is only completed at the screening appointment and administration of the BNT and JLO only occur at the baseline pre-treatment visit and the 12-months post-treatment follow up visit to minimize participant fatigue and familiarity with the test materials. Administration of the NCT at the screening visit will serve two purposes. Data obtained from the screening visit will ensure that subjects who are enrolled in the trial meet criteria for early AD based on the more comprehensive battery of tests, as diagnosis of dementia is improved with use of quantitative measurement of multiple domains. The NCT at this screening visit will also expose participants to the NCT and since practice effects are greatest between the first and second exposure to NCT, practice effects will be minimized using this exposure and repeated measures ANOVAs.

Psychological functioning and quality of life (QOL) will also be evaluated to monitor participants' emotional status throughout the trial. The Patient Health Questionnaire-9 and the Generalized Anxiety Disorder-7 questionnaires will be used to assess depression and anxiety, respectively. If any participant endorses suicidal ideation on the PHQ-9, the Suicide Behaviors Questionnaire-Revised (SBQ-R) will be administered to fully evaluate the participant's suicidal ideation and study stopping rules will be implemented as needed to ensure the individual's safety. QOL will be evaluated by the Quality of Life in Alzheimer's disease (QOL-AD) and Quality of Life in Late-stage Dementia (QUALID) and Everyday Cognition (ECog) questionnaires (patient and caregiver forms).

Concern may be raised regarding the use of whole brain irradiation and its potential deleterious effect on neurocognitive testing. There have been reports on post-radiation neurocognitive testing in the setting of prophylactic cranial irradiation (PCI), which is whole brain fractionated RT commonly employed for patients with pulmonary small cell carcinoma. The standard whole brain PCI dose is 2.5 Gy x 10, considerably higher than the 2.0 Gy x 5 or 2.0 Gy x 10 schemes planned in the present study. Furthermore, patients in the PCI studies also received chemotherapy in addition to whole brain irradiation, and chemotherapy itself effects long-term NCF. In these PCI reports, if any neurocognitive decline was identified, it was modest, occurred within a short interval, e.g. 6-9 months, and improved. The investigators are thus proposing a 9-month follow up period for the 1st subject cohort (2.0 Gy x 5) before proceeding with the 2nd cohort (2.0 Gy x 10), although both cohorts will undergo NCF and QOL testing through 12 months.

Grosshans and colleagues from M. D. Anderson found that PCI is "unlikely to significantly affect NCF." They evaluated cognitive function in small cell lung cancer patients who received PCI (mean 2.5 Gy x 10). After chemotherapy, but before PCI, 47% already had evidence of impaired cognitive function. On multivariate analysis, there were no significant further declines after PCI. On univariate analysis, there were unsustained, early decreases in executive and language function, which did not persist with follow-up. A Japanese group applied the Hopkins Verbal Learning Test (revised Japanese version, HVLT-R) in 40 whole brain RT patients, at baseline, 4 months, and 8 months. Whole brain fractionation was either 2.5 Gy x 4, 3.0 Gy x 10, or 2.5 Gy x 10. The respective probabilities of decline in HVLT-R total recall at 4 months were, respectively, 40%, 7%, and 0%, and at 8 months 13%, 14% and 0% (48).

Also applicable is a recent report of whole brain (and whole spine) RT for medulloblastoma in children, a population believed more vulnerable to cognitive decline from RT. They did not receive chemotherapy, rather RT alone, 36 Gy in 36 fractions (1.0 Gy BID) to the entire brain and spine, followed by a boost to 68 Gy in 68 fractions to the tumor bed, typically posterior fossa. Using the Wechsler Intelligence Scale for Children to give verbal quotient, performance quotient, and full-scale intelligence quotient, cognitive function was preserved for all test domains throughout the study at 3 months, 1 year, and 2 years, with no decline over time.

Low dose whole brain RT has demonstrated safety in many studies, and the investigators will be using even lower doses. These lower radiation therapy doses have a history of excellent success for patients with non-cerebral amyloidosis, and have had durable response combined with the necropsy / neurocognitive testing in genetically altered Alzheimer's disease mouse model, the investigators decided to proceed with a human trial, using fractionated whole brain radiation doses of 2.0 Gy x 5, then 2.0 Gy x 10. Subjects will be followed with neurocognitive testing at 6 weeks, 3, 9 and 12 months post RT. Additionally, given that the development of supranuclear cataract has been reported in a high percent of AD patients, the investigators will recommend ocular testing at baseline and at 1 year to assess a potential abscopal effect, collateral benefit to the non-targeted lenses from treatment of the primary disease in the brain.

With respect to the development of cataracts in association with AD, early and accurate diagnosis of Alzheimer's disease (AD) is still a challenge and the confirmatory diagnosis is made by presence of features including beta-amyloid plaques postmortem. In 2014, Tian et al suggested that AD may have a common pathophysiology with supranuclear deposits of beta-amyloid in the human lens. The brain and the lens tissue both arise from the ectoderm tissue (neuroectoderm and surface ectoderm respectively). Their conclusions were based on a meta-analysis of studies, which provided mixed data regarding the correlation of beta-amyloid in the lens samples of patients with AD, Down syndrome and controls. Given the chronicity of the terminally differentiated cell types in the lens that may be affected by Alzheimer disease's pathology, they concluded that there is a possibility than an ocular biomarker for early AD may exist in the lens. This would suggest that an early ophthalmic examination may provide a window of hope into early diagnosis of AD. It may also provide an opportunity for early treatment and perhaps monitoring of improvement in supranuclear cataracts with systemic therapy.

A precedent for this is already found in Wilson's disease. Kayser-Fleischer (K-F) ring seen in Wilson's disease (WD) is due to copper deposition in the Descemet's membrane in the sclero-corneal junction in the eye. Although believed to be pathognomic of WD, it may be seen in many other hepatic conditions and intraocular copper-containing foreign bodies. The K-F ring detected in pre-symptomatic cases of WD may lead to speedy diagnosis and early management. Co-relation of K-F ring in WD to the disease severity, disappearance with successful treatment, reappearance with non-compliant treatment aids in management of WD. K-F ring detection in first-degree relatives of the index case is also important.

With the proposed ocular exams at baseline and at 9-months post treatment, the investigators hope to detect any cataracts in the subjects and effects of the proposed radiation treatments. The questions the investigators will have are how often they encounter them in early Alzheimer's and whether they improve (an abscopal effect) after radiation therapy, even though the lenses will be excluded from the RT treatment fields. Exams will only be done for subjects who have at least one natural lense still present. Subjects with previous cataract corrections will not have ocular exams performed.

ELIGIBILITY:
Inclusion Criteria:

* Must be a native English speaker with a LAR available for consenting.
* Able to complete neurocognitive function assessments, psychological function assessments, and QOL assessments administered at screening visit.
* Rosen Modified Hachinski Ischemic Score less than or equal to 4
* Estimated Survival of greater than 12 months
* Meets the clinical definition of AD based on NINCDS-ADRDA criteria, with confirmatory F-2-DG and F-Florbetapir (Amyvid) PET scan findings
* If on any of the following medications, must be on a stable dose for 60 days or greater: Rivastigmine, Donepezil, Memantine, Glantamine, Tacrine.

Exclusion Criteria:

* Current or past history of any oncologic disease mitigating low dose whole brain RT
* Evidence of substance abuse (Alcohol/or other drugs or dependences during previous 12 months (DSM-V criteria)
* Clinically or radiographically significant evidence of stroke
* Evidence of subdural hygromas or subdural hematomas
* Active or recent (defined as within 3 months of screening) cerebral infection or hemorrhage
* Any current conditions that may lead to the subject being in an immuno-compromised state
* Any previous history of cranial radiation
* History of seizure activity
* History of Hydrocephalus
* Evidence of active dermatological skin disease of the scalp (except Actinic Keratosis)
* Evidence of clinically significant major depressive disorder identified in a psychological diagnostic interview according to the criteria of the Diagnostic and Statistical Manual of Mental Disorder, Fifth Edition (DSM-V)
* Evidence of psychotic disorder or psychotic episode or bipolar affective disorder identified in a psychological diagnostic interview according to the criteria of the Diagnostic and Statistical Manual of Mental Disorder, Fifth Edition (DSM-V)
* Evidence of active suicidal or homicidal ideation according to psychological diagnostic interview
* Currently receiving other experimental treatments
* Currently requiring full-time institutional care

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-05; Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Harris, M.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Rogers CL, Lageman SK, Fontanesi J, Wilson GD, Boling PA, Bansal S, Karis JP, Sabbagh M, Mehta MP, Harris TJ. Low-Dose Whole Brain Radiation Therapy for Alzheimer's Dementia: Results From a Pilot Trial in Humans. Int J Radiat Oncol Biol Phys. 2023 Sep 1;117(1):87-95. doi: 10.1016/j.ijrobp.2023.03.044. Epub 2023 Mar 18. PMID 36935024

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects 1-15: 10 GY in 5 daily fractions: Subjects 1-15 10 GY in 5 daily fractions
- Subjects 16 - 30: 20 GY in 10 daily fractions: Subjects 16-30 20 GY in 10 daily fractions
Period: Overall Study
Arm/Group | Subjects 1-15 | Subjects 16 - 30
Started | 5 | 0
Completed | 5 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in the second arm. The first 15 participants were to be assigned to the first arm and the study was terminated after enrolling only 5 participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects 1-15 | Subjects 16 - 30 | Total
Number analyzed (Participants) | 5 | 0 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 5 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 0 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 |  | 5

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Toxicity Associated With Delivery of Low Dose Fractionated Whole Brain Irradiation in Subjects With Early Alzheimer's Dementia According to ADRDA Criteria.
Description: Evaluate the toxicity associated with the delivery of low dose fractionated whole brain irradiation in subjects with early Alzheimer's dementia using the CTCAE toxicity grading system. The scale is 0 - 5 with 0 being no toxicity and 5 being fatal.
Time Frame: 48 months
Measure: Median (Full Range); unit: grade of toxicity
Arm/Group | Subjects 1-15
Number analyzed (Participants) | 5
grade of toxicity
  Skin toxicity | 2 [0 to 2]
  Eye toxicity | 0 [0 to 2]
  Ear toxicity | 0 [0 to 2]
  Central Nervous System toxicity | 2 [2 to 3]
  Other toxicity | 1 [0 to 2]

2. Secondary Outcome: Neurocognitive Function: Verbal Learning and Memory
Description: Patients will complete the Hopkins Verbal Learning Test-Revised (HVLT-R) which is a paper and pencil assessment. Overall scores will be reported. Scores range from 0 to 26 with higher scores indicating better functioning.
Time Frame: Baseline to 12 months
Population: Due to low power because of the small number of participants enrolled, change scores have not been calculated. Baseline and 12 month median scores and ranges are reported.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Subjects 1-15
Number analyzed (Participants) | 5
score on a scale
  Baseline | 18 [8 to 21]
  12 months | 15 [4 to 20]

3. Secondary Outcome: Neurocognitive Function: Visuospatial Memory
Description: Patients will complete the Brief Visuospatial Memory Test-revised which is a paper and pencil assessment. Overall scores will be reported. Scores range from 0 to 36 with higher scores indicating better functioning.
Time Frame: Baseline to 12 months
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Subjects 1-15
Number analyzed (Participants) | 5
score on a scale
  Baseline | 12 [5 to 17]
  12 months | 10 [4 to 22]

4. Secondary Outcome: Neurocognitive Function: Cognitive Function
Description: Patients will complete the Mini-Mental State Exam (MMSE) which is an interview style assessment. Overall scores will be reported. Scores range from 0 to 30 with higher scores indicating better functioning.
Time Frame: Baseline to 12 months
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Subjects 1-15
Number analyzed (Participants) | 5
score on a scale
  Baseline | 25 [22 to 25]
  12 months | 26 [13 to 29]

5. Secondary Outcome: Psychological Functioning: Depression
Description: Patients will complete the PHQ-9 (Patient Health Questionnaire-9) which is an interview style assessment. Overall scores will be reported. Scores range from 0 to 27 with lower scores indicting lower depression.
Time Frame: Baseline to 12 months
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Subjects 1-15
Number analyzed (Participants) | 5
score on a scale
  Baseline | 2 [0 to 2]
  12 Months | 3 [1 to 8]

6. Secondary Outcome: Psychological Functioning: Anxiety
Description: Patients will complete the GAD-7 (General Anxiety Disorder-7) which is an interview style assessment. Overall scores will be reported. Scores range from 0 to 21 with lower scores indicating lower levels of anxiety.
Time Frame: Baseline to 12 months
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Subjects 1-15
Number analyzed (Participants) | 5
score on a scale
  Baseline | 3 [1 to 3]
  12 Months | 1 [0 to 6]

7. Secondary Outcome: Quality of Life in Alzheimer's Disease
Description: Patients will complete the Quality of Life in Alzheimer's Disease (QOL-AD) which is an interview style assessment. The QOL-AD is a 13-item questionnaire designed to provide both a patient and a caregiver report of the quality of life (QOL) for patients who have been diagnosed with Alzheimer Disease. Overall scores will be reported. Scores range from 13 to 52 with higher scores indicating better quality of life.
Time Frame: Baseline to 12 months
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Subjects 1-15
Number analyzed (Participants) | 5
score on a scale
  Baseline | 46 [34 to 46]
  12 Months | 40 [39 to 46]

8. Secondary Outcome: Cognitive and Functional Decline
Description: Patients will complete the Everyday Cognition (ECog) which is an interview style assessment. Overall scores will be reported. Scores range from 39 to 156 with lower scores indicating less decline in cognition.
Time Frame: Baseline to 12 months
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Subjects 1-15
Number analyzed (Participants) | 5
score on a scale
  Baseline | 66 [45 to 72]
  12 Months | 64 [32 to 88]

ADVERSE EVENTS:
Time Frame: 48 months
Arm/Group | Subjects 1-15
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/00/NCT02769000/Prot_SAP_000.pdf